CLINICAL TRIAL: NCT00523536
Title: Latinos Using Cardio Health Actions to Reduce Risk (LUCHAR): Evaluation of a Navigator-Nurse Care Team on Hypertension and Cardiovascular Disease Risk
Brief Title: Evaluation of a Navigator-Nurse Care Team on the Management of High Blood Pressure and Cardiovascular Disease Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Ed Havranek, Physician, Denver Health and Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 486; U01HL079160 (NIH); U01HL079160-03 (NIH)
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2009-04

CONDITIONS: Hypertension
Keywords: High Blood Pressure; Cardiovascular
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patient navigator-nurse disease management intervention
  Interventions: Behavioral: Patient Navigator - Nurse Team Intervention
- 2 (No Intervention): Usual clinical care

INTERVENTIONS:
Behavioral: Patient Navigator - Nurse Team Intervention — The patient navigator-nurse disease management intervention for treating hypertension and its associated cardiovascular risk factors will use information obtained in earlier phases of the LUCHAR grant: i.e., algorithms, risk factor profiles, and qualitative data from focus groups and interviews. The study will test the effect of this intervention on blood pressure control and utilization of hospital services in adult patients with hypertension.
  Arms: 1

SUMMARY:
The purpose of this trial is to study the effect of a patient navigator-nurse team in improving the management of hypertension and other cardiovascular disease risk factors in a health care system taking care of a vulnerable, mostly Latino population.

DETAILED DESCRIPTION:
This study represents one phase of a large partnership grant with The Colorado Health Outcomes Program of the University of Colorado at Denver Health Sciences Center (UCDHSC) and Denver Health and Hospital Authority (DH). The overarching goal of Latinos Using Cardio Health Actions to Reduce Risk (LUCHAR) is to improve the primary and secondary prevention of cardiovascular disease (CVD) in Hispanics through a comprehensive research program aimed at (1) increasing awareness of CVD risk in the Hispanic community and increasing participation of high risk Hispanics in the health care system, (2) developing more effective models of care delivery for high risk patients in a health system, and (3) identifying markers that will more effectively identify Hispanic patients at high risk of CVD than current approaches based on traditional risk factors.

This trial has been designed to assess the effectiveness of a quality improvement project which focuses on the hypertensive multiracial underserved population within the Denver Health system. In addition, we are hoping at study end to have developed and validate this project as an efficient and sustainable approach to improving blood pressure control and controlling cardiovascular risk factors, especially in the vulnerable patient population served at Denver Health.

The objective of this quality improvement program is to conduct a randomized, primary care-based, efficacy trial evaluating the effectiveness of a patient navigator-nurse disease management intervention for treating hypertension and its associated cardiovascular risk factors using information obtained in earlier phases of the LUCHAR grant: i.e., algorithms, risk factor profiles, and qualitative data from focus groups and interviews. The study is designed to test the hypothesis that a patient navigator-nurse assisted intervention will improve blood pressure (BP) in vulnerable hypertensive patients, compared with usual clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Active patients from the Target Adult Health Clinic
* Identified with a diagnosis of hypertension
* Uncontrolled hypertension (2 of 3 last BP measurements above target BP range; target BP is defined at 140/90 or 130/80 mm Hg for people with diabetes or kidney disease)

Exclusion Criteria:

* Pregnant or breastfeeding
* End-stage kidney disease requiring dialysis
* Co-morbid illness with life expectancy less than 12 months
* Institutionalized individuals because of the potentially confounding factors due to severe co-morbidity or other medical conditions

Ages: 21 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2007-05; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Change in SBP level | Measured at Year 1

SECONDARY OUTCOMES:
Percentage of participants with BP control by JNC-7 guidelines, adherence with BP medications, lipid control, change of HgbA1c for participants with diabetes, and change in smoking status/BMI | Measured at Year 1
Utilization of urgent care visits/emergency department/hospitalizations | Measured at Year 1

CONTACTS AND LOCATIONS:
Overall Officials: Raymond O. Estacio, MD, Principal Investigator — Denver Health, University of Colorado at Denver Health Sciences Center
Locations (1):
- East Adult Clinic, Denver Health, Denver, Colorado, United States